CLINICAL TRIAL: NCT06921980
Title: Brain Function and Psychological Assessment in Patients With Autoimmune Hemolytic Anemia Undergoing Cell Therapy
Brief Title: Brain Function and Psychological Changes Related to Cell Therapy for Autoimmune Hemolytic Anemia
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tianjin University (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2025011
Record Dates: First submitted 2025-04-02; First posted 2025-04-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-04

CONDITIONS: CAR T-cell Therapy; Autoimmune Hemolytic Anemia; Brain Function; Psychological Well-Being
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental: Brain function and psychological changes in AIHA patients will be monitored throughout cell therapy.
  Interventions: Other: Brain function and psychological assessment

INTERVENTIONS:
Other: Brain function and psychological assessment — Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.

SUMMARY:
Cell therapy is an innovative treatment with significant efficacy in hematologic and certain autoimmune diseases. Although it offers potential benefits for autoimmune hemolytic anemia (AIHA), it may result in cognitive and other potential impairments, which can adversely affect patients' cognition and behavior.

Brain function and psychological assessment are essential for the early detection of potential impairments, allowing timely interventions to prevent complications and ensure patient safety. This study aims to comprehensively evaluate the physical and psychological impacts of cell therapy on AIHA patients to develop safer and more effective treatment strategies that enhance their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIHA
* Subjects will receive cell therapy such as CAR T-cell therapy
* Male or female, aged 18-65 years
* Willing and able to comply with the requirements for this study and written informed consent

Exclusion Criteria:

* History of psychiatric illness
* History of severe brain disease
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/refractory AIHA who will receive cell therapy, such as CAR T-cell therapy, from 2025 to 2026.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration changes in oxygenated hemoglobin (HbO) and de-oxygenated hemoglobin (HbR) | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  Functional Near Infrared Spectroscopy (fNIRS) is a non-invasive brain imaging modality, that can be used to measure HbO and HbR concentrations.
Psychological change | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  The Big Five Inventory-2(BFI-2) is used to measure the five broad dimensions of personality: openness, conscientiousness, extraversion, agreeableness, neuroticism. Higher scores indicate a stronger presence of that personality trait.
Anxiety symptoms | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  Hamilton anxiety scale(HAMA) is used to examine anxiety in AIHA patients, with higher total scores indicate more severe anxiety symptoms. The total score range is 0-56.
Depression symptoms | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  Hamilton depression scale(HAMD) is used to examine depression in AIHA patients, with higher total scores indicate more severe depression symptoms. The total score range is 0-52.

SECONDARY OUTCOMES:
Sleep quality | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality, with a higher global score indicating poorer sleep quality. The global score range is 0-21.
Physical fatigue | Patients will be assessed before cell therapy and on Days 1, 4, 7, 10, 14, 21, and 28 after treatment.
  It measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale. The total possible score is 0-52 points, with higher scores indicating less fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No